CLINICAL TRIAL: NCT05661799
Title: Psychological Levers of Commitment and Persistence in Physical Activity in People With Type 2 Diabetes. PerPA2Temps Study
Brief Title: Persistence of Physical Activity in People With Type 2 Diabetes Over Time.
Acronym: PerPA2Temps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Siel Bleu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PerPA2Temps
Record Dates: First submitted 2022-11-09; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Diabetes Mellitus, Type 2; Physical Activity; Psychological
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The proposed intervention consists of one hour of adapted physical activity per week for 12 weeks, led by a professional. In addition to this intervention, the intervention includes two 15-minute sessions, one before and one after the session. At the end of each session, a PA challenge and a positive reinforcement exercise will be proposed. The participants will have a week to try to achieve these. In addition to these two 15-minute sessions, participants will benefit from a one-and-a-half hour group session for information and experience sharing. The aim of this session is to discuss different topics related to diabetes.
  Interventions: Behavioral: Intervention Group
- Control group (Active Comparator): The proposed intervention consists of one hour of adapted physical activity per week for 12 weeks, led by a professional.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Intervention Group — The programme is a PA programme consisting of one weekly session for 12 weeks. The one hour of PA is supplemented by two 15-minute periods. At the end of each session, a PA challenge and a positive reinforcement exercise are proposed for the coming week. At the beginning of the next session, the facilitator has a dedicated time to give feedback on these challenges (successes and difficulties encountered). At the end of each session, the facilitator explains the theme of the next challenge and exercise. For the challenge, three options are proposed. Each participant chooses the option he/she prefers. Positive reinforcement exercises are also offered in the same way. They aim to strengthen motivation, hope and the sense of self-efficacy (SEP). In addition to these two 15-minute sessions, participants are offered a one-and-a-half hour group session for information and experience sharing. The aim of this session is to discuss different themes.
  Arms: Intervention Group
Behavioral: Control Group — The programme is a PA programme consisting of one weekly session for 12 weeks.
  Arms: Control group

SUMMARY:
Many programmes exist to enable patients to engage in physical activity, but it is clear that the objectives are often not achieved in terms of quality, quantity or intensity of practice. In this study, the aim is to find alternatives, assuming that strengthening patients' self-efficacy, meeting their basic needs and increasing their level of hope will have an impact on their motivation to practice, which in turn will have an impact on their actual practice. The aim is to develop and implement an innovative intervention programme and to identify the interactions between the variables that are assumed to predict engagement in practice.

DETAILED DESCRIPTION:
Type 2 diabetes is one of the chronic pathologies that can be treated, in part or in full, by respecting hygienic-dietary rules (i.e. recommendations on dietary balance and physical activity). Numerous studies have demonstrated the benefits of physical activity (Duclos et al., 2012; Sigal et al., 2013) but few patients change their behaviour over the long term. A field of psychology has put forward certain notions that can be levers for practice: the theory of hope, the feeling of personal efficacy (SEP), motivation and basic psychological needs. Some motivational programmes for physical activity (PA) have been developed on the basis of these concepts in different fields (i.e. work, school) but, to our knowledge, in France, none has yet been developed in the field of health and a fortiori in the management of people with diabetes.

The main objective of this study is to develop and implement an innovative motivational intervention programme in adapted physical activity (APA) for type 2 diabetic patients (T2DM). The aim of this programme is to enable them to improve their chances of engagement and persistence in physical activity. To this end, the investigators would like to study the effect of this type of programme on physical activity.

Secondly, the investigators would like to study, on the one hand, the evolution and the interactions between the different psychological variables in the framework of this innovative intervention programme. On the other hand, the investigators want to study the impact of the intervention on physical fitness, commitment and satisfaction with physical activity.

The study will be set up within the framework of the APA sessions provided by the Siel Bleu association. The subjects will be new exercisers, type 2 diabetics not treated with insulin, having been included through the various partners of Siel Bleu.

the investigators will have an intervention group and a control group. The control group will benefit from a standard APA programme offered by Siel Bleu. A standard APA programme consists of one-hour sessions in a group of up to 15 people. The objective of these Siel Bleu programmes is to maintain or improve the physical capacities of the participants. To achieve this, several session themes are addressed (i.e. endurance, muscular strength of upper and lower limbs, balance, flexibility, coordination). The intervention group will participate in this APA programme with an information and experience sharing session as well as APA challenges and various positive reinforcement exercises. Data will be collected in the form of questionnaires at inclusion, at the end of the programme and at 3, 6 and 12 months after the programme.

For this study, with a risk α=5%, a guaranteed power of 80%, a delta of 25% and a standard deviation of 22.5 minutes, the investigators will need 298 subjects equally distributed in the two groups.

Our primary endpoint will be the amount of physical activity. This will be measured by the Global Physical Activity Questionnaire (GPAQ), which will allow us to differentiate between the various intensities of physical activity and the contexts in which it is performed.

Thanks to our innovative physical activity programme combining weekly PA practice with PA challenges and positive reinforcement exercises, the investigators expect an increase in the amount of physical activity, 12 months after the programme, twice as high as in the control group. We also expect to see changes in feelings of self-efficacy (SEP) and levels of trait and state hope as well as more self-determined motivation.

The investigators also hope that the results will allow us to determine the statistical power of the correlations between the variables as well as to identify typical profiles to predict the evolution of the amount of physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Subject over 18 years of age
* Subject who has given signed consent to participate in the protocol
* Type 2 diabetic subject not treated with insulin
* Subject participating for the first time in adapted physical activity sessions provided by Siel Bleu
* Subject understanding and reading French

Exclusion Criteria:

* Subjects with major health problems that prevent them from continuing the programme.
* Subjects who have withdrawn their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Change in amount of physical activity assessed by the French Version of GPAQ | Pre-intervention/immediately after the intervention, at 3, 6 and 12 months after the intervention
  The evolution of the quantity of physical activity will be the main criterion of judgment. It will be measured by the Global Physical Activity Questionnaire, which will allow for differentiation of intensities and contexts of practice. This questionnaire will be administered at each evaluation time proposed by the study (before/after, at 3, 6 and 12 months). The higher the score (in Metabolic Equivalent of Task/minutes/weeks), the greater the amount and intensity of physical activity performed.
  The comparison between the pre- and post-programme assessments (e.g. T0 and T1) will allow the direct effect of the programme on the amount of physical activity to be determined. The other assessments (e.g. T2, T3 and T4) will determine the persistence of this practice over time.

SECONDARY OUTCOMES:
Change in the subjects' motivational profile towards a more self-determined motivation assessed by the French Version of the Motivation for Physical Activity for Health Scale | Pre-intervention/immediately after the intervention, at 3, 6 and 12 months after the intervention
  To assess the motivation of the subjects, the Motivation for Physical Activity for Health Scale will be used. It measures the quality of contextual motivation with three items per dimension (intrinsic motivation, integrated regulation, identified regulation, introjected regulation, external regulation and amotivation). Subjects will respond with a 7-point Likert scale ranging from 1 (does not match at all) to 7 (matches very strongly).
Change in the satisfaction of basic psychological needs assessed by the French Version of The Basic Psychological Needs. | Pre-intervention/immediately after the intervention, at 3, 6 and 12 months after the intervention
  The Basic Psychological Needs in Sport questionnaire assesses the three dimensions of basic psychological needs using five items per need: satisfaction of the need for autonomy (e.g., I feel free to make my own choices), satisfaction of the need for affiliation (e.g., I feel comfortable with others), and satisfaction of the need for competence (e.g., I feel successful). Subjects will respond using a Likert scale ranging from 1 (not at all true) to 7 (completely true). This questionnaire will be administered at each evaluation time proposed by the study.
Change in self-efficacy assessed by the French Version of The Self-Efficacy Questionnaire | Pre-intervention/immediately after the intervention, at 3, 6 and 12 months after the intervention
  The Self-Efficacy Questionnaire (SEP) is composed of 40 items corresponding to cognitive-emotional and behavioural conditions. These 40 items are divided into four categories, each based on 10 descriptors of SEP manifestations: management of eating behaviour, physical activity, body image and the gaze of others, and social relations. Subjects are asked to respond on a Likert-type scale ranging from 0 to 10 and to indicate a score out of 10 from "not at all capable" to "very capable". This score yields five scores; one for each difficulty, calculated over 10 items. An overall score is calculated out of 40.
Change of initial state hope level assessed by the French Version of the State Hope Scale | Pre-intervention/immediately after the intervention, at 3, 6 and 12 months after the intervention
  The level of state hope is measured by a self-administered questionnaire. In this questionnaire, the total hope score is calculated using six items, three of which correspond to the motivational component and three to the operative component. Responses to these items are based on a six-point Likert-type scale, ranging from 1 (Strongly disagree) to 6 (Strongly agree). The total state expectancy score will be evaluated on 36 points. The operant and motivational component sub-scores will be assessed on 18 points each.
Change in dispositional hope level assessed by the French Version of the Adult Dispositional Hope Scale | Pre-intervention/immediately after the intervention
  This self-evaluation scale is composed of 12 items corresponding to three different categories: the operative component includes four items, the motivational component also includes four items, and the remaining four items are decoys. Subjects will be able to respond to the questions using a Likert scale ranging from 1 (Always false) to 8 (Always true). The total dispositional hope score will be between 8 and 64 points. The operant and motivational component subscores will range from 4 to 32 points each.
Change in dispositional optimism level assessed by the French Version of The Life Orientation Test-Revised | Pre-intervention/immediately after the intervention
  The Life Orientation Test-Revised is composed of 10 items corresponding to three categories: positive expectations associated with three items, negative expectations represented by three items, and the other four items corresponding to decoys. The subjects will answer the questionnaires on their own using a Likert scale ranging from 0 (Totally Disagree) to 4 (Totally Agree). This questionnaire provides an overall optimism score as well as two sub-scores corresponding to positive and negative expectations.
Change in physical condition assessed by The 6-Minute Walk Test | Pre-intervention/immediately after the intervention
  The 6-Minute Walk Test is a standardised test to measure exercise capacity in an objective way. In this test, the subject is asked to walk as far as possible for six minutes. Several data are then collected: distance covered (in metres), oxygen saturation, heart rate (in beats per minute) and degree of breathlessness (on a Borg scale ranging from 1 to 10). For our study, heart rate (HR) and degree of breathlessness will be collected before the test, just after and one minute after the end of the test. During the test, the subject will be kept informed of the time remaining every minute. At the same time, the subject will receive encouragement (i.e. "That's very good, keep it up").
Subject attendance assessed by an attendance grid | Through intervention completion, that is, 12 weeks
  Completed by the facilitator, the number of participants at each session, attendance (presence or absence of each participant at each session), completion of active challenges and weekly positive reinforcement exercises is recorded.
Participant satisfaction assessed by a study-specific questionnaire | Immediately after the intervention
  The satisfaction questionnaire assesses different aspects of the programme. Questions about the physical activity sessions will be asked (i.e. satisfaction with the content, diversity, user-friendliness, etc.). Satisfaction with the facilitator will also be assessed (i.e. ability to adapt the exercises, to motivate the group, to promote autonomy, etc.). The benefits of the programme will be judged on the basis of various categories (i.e. physical, biological, psychological and social). Participants will have the opportunity to rate the programme on a scale of 1 to 10 (10 being the highest) and to leave various comments. For those who benefited from the specific programme under study, the questionnaire includes an additional module to assess satisfaction with the active challenges, the positive reinforcement exercises and the information and experience sharing group.
Individual demographic and socio-economic data assessed by a specific form for the study | Pre-intervention
  The subject completes an information sheet including: age, gender, level of education, socio-professional category, and place of residence.
Initial medical data assessed by a specific form for the study | Pre-intervention
  The subject completes an information sheet including: personal and family history and height (in centimetres)
Progressive medical data assessed by a specific form for the study | Pre-intervention/immediately after the intervention, at 3, 6 and 12 months after the intervention
  The subject completes an information sheet including: weight (in kilograms), treatment type and glycated haemoglobin (in %)

CONTACTS AND LOCATIONS:
Overall Officials: Elise Maudet-Coulomb, Ms, Principal Investigator — Université de Lorraine, EA 4360 APEMAC, Metz, France; Charles Martin-Krumm, PhD, Study Chair — Université de Lorraine, EA 4360 APEMAC, Metz, France; Jean-Christophe Mino, PhD, Study Chair — Institut de recherche Siel Bleu, Paris France
Locations (1):
- Elise Maudet-Coulomb, Angers, Maine Et Loire, France

IPD SHARING:
Plan to Share IPD: No